CLINICAL TRIAL: NCT01099410
Title: Apoptotic Cell Ingestion by Normal Human Alveolar Macrophages
Brief Title: Apoptotic Cell (AC) Uptake by Human Alveolar Macrophages (AM)
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Curtis 0015
Record Dates: First submitted 2010-03-30; First posted 2010-04-07 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: macrophages, alveolar; monocytes; Receptor Protein-Tyrosine Kinases; Humans; Phagocytosis; Lung; in vitro
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood, white blood cells, serum, bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: volunteer subjects
  Interventions: Procedure: Fiberoptic bronchoscopy; Procedure: blood draw; Procedure: intravenous catheter

INTERVENTIONS:
Procedure: Fiberoptic bronchoscopy — which a flexible video instrument is passed via the nose or mouth, through the vocal cords and into the lungs. During the procedure, portions of the lungs will be washed ("lavaged") with a salt water solution, to collect the alveolar macrophages. This procedure involves conscious sedation, so that a driver is required on the day of the bronchoscopy. The entire procedure, including placement of an intravenous line to administer medications, local anesthetics, the bronchoscopy itself, and the recovery period, takes about 2.5-3 hours.
Procedure: blood draw — Blood will be collected at the enrollment visit to test the subject to exclude disorders that would make it unsafe to perform the bronchoscopy, including severe anemia, infection, or disorders of kidney or liver function.
Procedure: intravenous catheter — An intravenous catheter is placed on the day of the bronchoscopy to permit administration of sedative medications.
  Other Names: IV

SUMMARY:
The purpose of this study is to compare the ability of two types of white blood cells to eat dead host cells, and how this process affects their ability to protect the body from infection. The two cell types are monocytes, a cell in the bloodstream, and alveolar macrophages, a cell in the lung that is ultimately derived from monocytes

DETAILED DESCRIPTION:
Volunteers, who may be Veterans or non-Veterans, will be screened by a series of questionnaires, chest X-ray, spirometry, EKG, blood work, and a complete history and physician examination by a study physician. Those who qualify for the study and agree via informed consent, will undergo a fiberoptic bronchoscopy on a separate day for the initial visit. Bronchoscopy is a procedure in which a flexible video instrument is passed via the nose or mouth, through the vocal cords and into the lungs. During the procedure, portions of the lungs will be washed ("lavaged") with a salt water solution, to collect the alveolar macrophages. This procedure involves conscious sedation, so that a driver is required on the day of the bronchoscopy. The entire procedure, including placement of an intravenous line to administer medications, local anesthetics, the bronchoscopy itself, and the recovery period, takes about 2.5-3 hours. The cells collected by bronchoscopy will be studied in the research laboratory, and used entirely in that procedure.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or non-Veteran
* Able to give informed consent

Exclusion Criteria:

* Unstable heart disease
* Other systemic disease and unlikely to survive at least 2 years
* Mental incompetence
* Prednisone >20 mg/day
* Participation in another interventional protocol within last 6 weeks
* Asthma
* Cystic fibrosis
* Clinically significant bronchiectasis
* Lung cancer or any cancer not in remission for at least 5 years
* Other inflammatory or fibrotic lung disease
* Use of antibiotics for a lung infection within the past 4 weeks
* Autoimmune disease, i.e., Rheumatoid arthritis, systemic lupus erythematosus, autoimmune hepatitis, Crohn's disease or other

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects recruited from the community; may be current or ex-smokers or never-smokers, but must be healthy enough to undergo research bronchoscopy safely.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
macrophage uptake of apoptotic cells in vitro | 1-7 days

SECONDARY OUTCOMES:
spirometric measurement of lung function | 1-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Curtis, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Bourdonnay E, Zaslona Z, Penke LR, Speth JM, Schneider DJ, Przybranowski S, Swanson JA, Mancuso P, Freeman CM, Curtis JL, Peters-Golden M. Transcellular delivery of vesicular SOCS proteins from macrophages to epithelial cells blunts inflammatory signaling. J Exp Med. 2015 May 4;212(5):729-42. doi: 10.1084/jem.20141675. Epub 2015 Apr 6. PMID 25847945
- [Result] Todt JC, Freeman CM, Brown JP, Sonstein J, Ames TM, McCubbrey AL, Martinez FJ, Chensue SW, Beck JM, Curtis JL. Smoking decreases the response of human lung macrophages to double-stranded RNA by reducing TLR3 expression. Respir Res. 2013 Mar 9;14(1):33. doi: 10.1186/1465-9921-14-33. PMID 23497334